CLINICAL TRIAL: NCT00029029
Title: RF Ablation of Painful Metastases Involving Bone
Brief Title: Radiofrequency Ablation in Relieving Pain in Patients With Bones Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Purpose: Supportive Care
Other Study IDs: CDR0000069180; RITA-201-00; MAYO-IRB-O-1223-00; MDA-ID-01534; RITA-IDE-G000177
Record Dates: First submitted 2002-01-04; First posted 2003-01-27 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Metastatic Cancer; Pain
Keywords: bone metastases; pain
MeSH Terms: conditions — Neoplasm Metastasis; Pain | interventions — Analgesia; Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: pain therapy
Procedure: radiofrequency ablation

SUMMARY:
RATIONALE: Radiofrequency ablation uses high-frequency electric current to kill tumor cells and may help to relieve pain caused by bone metastases.

PURPOSE: Phase II trial to study the effectiveness of radiofrequency ablation in relieving pain in patients who have bone metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of radiofrequency ablation, in terms of pain relief at 4 weeks, in patients with painful bone metastases.
* Determine the safety of this regimen in these patients.
* Compare the change in pain interference with daily life and analgesic use at 4 weeks vs baseline in patients treated with this regimen.
* Determine the time to recurrence of worst pain in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive radiofrequency ablation (RFA) to targeted tumor(s) on day 0 (multiple tumors may receive ablation in multiple sessions). Patients who achieve a reduction in worst pain of at least 2 points within 4-8 weeks but experience recurring pain at the RFA site or are diagnosed with a new painful lesion within 4-24 weeks receive 1 additional treatment to the recurring or new site.

Pain (using the Brief Pain Inventory scale of 0-10), analgesic use, and quality of life are assessed at baseline, on day 1, weekly for 4 weeks, and then every 2 weeks for 20 weeks.

Patients are followed for 6 months beyond the last RFA treatment.

PROJECTED ACCRUAL: A maximum of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed bone metastases
* Pain refractory to non-opioid analgesic medication and radiotherapy OR
* Patient is considered a poor candidate for opioid analgesics or radiotherapy
* Initial worst pain score within the past 24 hours at least 4 on a scale of 0-10
* Tumors deemed accessible for radiofrequency ablation
* No evidence of impending fracture in weight-bearing bones (more than 50% loss of cortical bone)
* Tumors must be more than 1 cm from critical structures including:

  * Spinal cord, brain, or other critical nerve structures
  * Large abdominal vessel (e.g., aorta or inferior vena cava)
  * Bowel or bladder

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Not specified

Life expectancy:

* More than 2 months

Hematopoietic:

* Platelet count at least 75,000/mm3

Hepatic:

* INR less than 1.5

Renal:

* Not specified

Other:

* Not pregnant or nursing
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 3 weeks since prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 3 weeks since prior radiotherapy

Surgery:

* Not specified

Other:

* At least 3 days since prior aspirin, ibuprofen, or other nonsteroidal anti-inflammatory drugs
* No concurrent anticoagulants

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-10-13 (Actual); Primary Completion 2002-10-24 (Actual); Study Completion 2002-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. William Charboneau, MD, Study Chair — Mayo Clinic
Locations (6):
- United States (6):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - St. Luke's Medical Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No